CLINICAL TRIAL: NCT01792050
Title: A Phase II Double-Blinded, Randomized, Placebo-Controlled Study of Indoximod in Combination With a Taxane Chemotherapy in Metastatic Breast Cancer
Brief Title: Study of Chemotherapy in Combination With IDO Inhibitor in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NLG2101
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Breast Cancer
Keywords: IDO; IDO Inhibitor; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; 1-methyltryptophan; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1A: Docetaxel + Placebo (Placebo Comparator): Arm 1A: Docetaxel 75 mg/m^2 IV given every 3 weeks (on day 8 of 21 day cycle), plus placebo PO BID (days 1-14 of 21 day cycle).
  Interventions: Drug: Docetaxel; Other: Placebo
- Arm 1B: Docetaxel + Indoximod (Experimental): Arm 1B: Docetaxel 75 mg/m^2 IV given every 3 weeks (on day 8 of 21 day cycle), plus Indoximod 1200 mg PO BID (days 1-14 of 21 day cycle).
  Interventions: Drug: Docetaxel; Drug: Indoximod
- Arm 2A: Paclitaxel + Placebo (Placebo Comparator): Arm 2A: Paclitaxel 80 mg/m^2 IV given weekly x3 followed by a week of rest (28 day cycle), plus placebo PO BID (days 1-21 of 28 day cycle).
  Interventions: Other: Placebo; Drug: Paclitaxel
- Arm 2B: Paclitaxel + Indoximod (Experimental): Arm 2B: Paclitaxel 80 mg/m^2 IV given weekly x3 followed by a week of rest (28 day cycle), plus Indoximod 1200 mg PO BID (days 1-21 of 28 day cycle).
  Interventions: Drug: Indoximod; Drug: Paclitaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel chemotherapy regimen given by vein over 1 hour on day 8 of each cycle.
  Other Names: Taxotere®
  Arms: Arm 1A: Docetaxel + Placebo; Arm 1B: Docetaxel + Indoximod
Other: Placebo — Placebo taken orally every morning 1 hour prior to breakfast and 1 hour prior to dinner on days 1-14. Six pills to be taken each time for a total of 12 pills per day.
  Arms: Arm 1A: Docetaxel + Placebo; Arm 2A: Paclitaxel + Placebo
Drug: Indoximod — Indoximod (1200 mg) taken orally every morning 1 hour prior to breakfast and 1 hour prior to dinner on days 1-14. Six 200 mg pills to be taken twice a day for a total of 12 pills per day.
  Other Names: 1-methyl-D-tryptophan, Indoximod, D-1MT, 1-MT
  Arms: Arm 1B: Docetaxel + Indoximod; Arm 2B: Paclitaxel + Indoximod
Drug: Paclitaxel — Paclitaxel chemotherapy regimen given by vein over 1 hour weekly x 3 followed by a week of rest each cycle.
  Other Names: Taxol
  Arms: Arm 2A: Paclitaxel + Placebo; Arm 2B: Paclitaxel + Indoximod

SUMMARY:
The purpose of this study is to compare the effects, good and/or bad, of standard of care therapy (docetaxel or paclitaxel) with or without the addition of 1-Methyl-D-tryptophan (referred to as indoximod) an experimental drug to find out which treatment is better.

DETAILED DESCRIPTION:
It is estimated that 232,340 US women will be diagnosed with and 40,030 women will die of breast cancer in 2013. Metastatic breast cancer is a terminal condition and treatments are palliative in nature. The median survival for patients with metastatic breast cancer is approximately 2.5 years. The standard therapies currently in use include anti-estrogen therapies (anastrazole, letrozole, fulvestrant, tamoxifen), chemotherapy agents (taxanes, capecitabine, navelbine, gemcitabine, eribulin, ixabepilone), targeted therapies (trastuzumab, lapatinib), and supportive care agents (zolendronic acid, denosumab). While breast cancer typically responds well to treatment, the response is transient and their disease becomes more refractory with continued therapy. Also, quality of life is a significant issue for these patients as many of these therapies are associated with significant side effects. Well tolerated, novel agents which improve the efficacy of existing chemotherapy agents would prove quite useful in managing metastatic breast cancer.

Preclinical data derived from MMTV-Neu mice with autochthonous tumors studied the interaction between indoximod and various chemotherapeutic agents. Mice with 5-10mm tumors were enrolled into control and treatment groups. Mice were treated with indoximod alone, chemotherapy alone (paclitaxel, doxorubicin, cyclophosphamide, and others), and the combination of indoximod and chemotherapy. treatment with indoximod or paclitaxel alone caused retardation of tumor growth in this model but no regressions were seen. the combination of indoximod plus paclitaxel caused 30% tumor regression and histologically there was significantly enhanced tumor cell death with the combination versus either agent alone. This synergism was abrogated when the mice underwent CD4+ T cell depletion prior to treatment with the combination, suggesting the immune response played a role in the observed effect. Based on this data and other reports suggesting systemic immunomodulating drugs like indoximod can synergize with chemotherapy agents such as taxanes, the decision was made to devise this combination of therapy of docetaxel or paclitaxel with indoximod in metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed estrogen/progesterone receptors (ER/PR) +/-; human epidermal growth factor receptor 2 (HER2)-, metastatic breast cancer.
* Metastatic disease that is evaluable on imaging. May have measureable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. Patients can also have non-measurable disease including bone only metastatic disease, evaluated by bone scan, PET or MRI.
* Any number of prior endocrine therapies in the metastatic setting are allowed. The patient must not have received any prior chemotherapy agents in the metastatic setting. Prior treatment with adjuvant docetaxel or paclitaxel is allowed if disease relapse occurred greater than 12 months from the completion of adjuvant therapy.
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1 (Karnofsky ≥60%).
* Life expectancy of greater than 4 months.
* Patients must have normal organ and marrow function as defined below: leukocytes ≥3,000/mcL, absolute neutrophil count ≥1,500/mcL, platelets ≥100,000/mcL, total bilirubin within normal institutional limits, aspartate aminotransferase AST(SGOT)/ alanine aminotransferase ALT(SGPT) ≤2.5 X institutional upper limit of normal, creatinine within normal institutional limits OR creatinine clearance ≥60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
* Patients with known brain metastases will only be eligible after their tumors have been treated with definitive resection and/or radiotherapy and they are neurologically stable for at least 1 month off steroids.
* Male and female subjects of child producing potential must agree to use adequate forms of contraception or avoidance of pregnancy measures prior to study entry, while enrolled on study and for a minimum of one month after completion of the study.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy for the treatment of metastatic breast cancer are not eligible. Patients who have had radiotherapy within 3 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier are not eligible.
* Patients who are currently receiving any other investigational agents.
* Patients with known active, untreated brain metastases should be excluded from this clinical trial. Those with previously treated inactive brain metastases with no evidence of active disease documented on brain MRI at least 4 weeks after radiation and off all steroids may be eligible.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel or tryptophan containing substances. This would include L-tryptophan or 5-hydroxy-tryptophan supplements. Also patients with a history of severe hypersensitivity reactions to docetaxel or to other drugs formulated with polysorbate 80 are excluded.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because indoximod is an immunoregulatory agent with the potential for abortifacient effects due to fetal rejection by the maternal immune system. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with indoximod, breastfeeding should be discontinued if the mother is treated with indoximod. Also, docetaxel and paclitaxel are category D cytotoxic agents and are not administered to pregnant females.
* Known HIV-positive patients and those with other acquired/inherited immunodeficiencies are ineligible due to the possibility of affecting the response to indoximod and the higher risk of active opportunistic infections.
* Patients with more than one active malignancy at the time of enrollment.
* Patients who have received any prior experimental active immunotherapy consisting of targeted monoclonal antibodies (ipilimumab) or pharmaceutical compounds are excluded.
* Patients with any active autoimmune disease (i.e. psoriasis, extensive atopic dermatitis, asthma, inflammatory bowel disease (IBD), multiple sclerosis (M.S.), uveitis, vasculitis), chronic inflammatory condition, or any condition requiring concurrent use of any systemic immunosuppressants or steroids for any reason would be excluded from the study. Any patient with an allo-transplant of any kind would be excluded as well. This would include those with a xenograft heart valve to avoid the potential risk of any immune reaction causing valvular degeneration. Mild-intermittent asthma requiring only occasional beta-agonist inhaler use or mild localized eczema will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2013-02; Primary Completion 2016-07-01 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 12 months
  The primary objective of this phase 2 study is the progression free survival of docetaxel or paclitaxel in combination with indoximod compared to docetaxel or paclitaxel plus placebo in metastatic breast cancer.

SECONDARY OUTCOMES:
Frequency and grade of adverse events of docetaxel and paclitaxel in combination with indoximod versus docetaxel alone | 12 months
  A secondary objective of this phase 2 study is to determine the safety/toxicity (frequency and grade of adverse events) of docetaxel or paclitaxel in combination with indoximod versus docetaxel or paclitaxel plus placebo.
Correlation of clinical and pathologic variables and clinical benefit (progression free survival rate) from treatment | 12 months
  A secondary objective of this phase 2 study is determining the correlation between clinical and pathologic variables and clinical benefit from docetaxel or paclitaxel and indoximod.
Median Overall Survival | 12 months
  A secondary objective of this phase 2 study is to observe median overall survival of all patients.
Objective Response Rate (Complete Response + Partial Response) | 12 Months
  A secondary objective is to determine the objective response rate (CR+PR) as measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) of docetaxel or paclitaxel + indoximod compared to docetaxel or paclitaxel plus placebo.

CONTACTS AND LOCATIONS:
Locations (39):
- United States (28):
  - University of Florida Health Cancer Center, Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Space Coast Cancer Center, Titusville, Florida
  - Cleveland Clinic - Florida, Weston, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Eastchester Center for Cancer Care, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest Baptist Hospital, Winston-Salem, North Carolina
  - Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic - Taussig Cancer Center, Cleveland, Ohio
  - Taussig Cancer Institute, Mayfield Heights, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Pennsylvania State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Paoli Hospital, Paoli, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Lynchburg Hematology Oncology, Lynchburg, Virginia
  - Peninsula Cancer Center, Newport News, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Wheaton Franciscan Healthcare- Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Baycare, Green Bay, Wisconsin
- Poland (11):
  - Research SiteR, Brzozów
  - Reserach Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Gorzów Wielkopolski
  - Reserach Site, Konin
  - Research Site, Krakow
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Rybnik
  - Research Site, Rzeszów
  - Research Site, Warsaw

REFERENCES:
- [Derived] Mariotti V, Han H, Ismail-Khan R, Tang SC, Dillon P, Montero AJ, Poklepovic A, Melin S, Ibrahim NK, Kennedy E, Vahanian N, Link C, Tennant L, Schuster S, Smith C, Danciu O, Gilman P, Soliman H. Effect of Taxane Chemotherapy With or Without Indoximod in Metastatic Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2021 Jan 1;7(1):61-69. doi: 10.1001/jamaoncol.2020.5572. PMID 33151286